CLINICAL TRIAL: NCT03570567
Title: Clinical Luminal Endoscopic Assessment of a Novel Suction (CLEANS) Technique for the Treatment of Esophageal Food Impaction
Brief Title: CLEANS Technique for the Treatment of Esophageal Food Impaction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Biomerics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M015-3-01
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Esophageal Food Impaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Piranha Treatment (Other): The food impaction will be treated using the Piranha endoscopic device.
  Interventions: Device: Piranha Treatment

INTERVENTIONS:
Device: Piranha Treatment — The piranha device is used with an endoscope to breakup/dislodge the food bolus.

SUMMARY:
This clinical investigation is to evaluate the safety, performance, and efficacy of a novel endoscopic technique for resolving esophageal food impactions by using a novel hollow suction catheter, Piranha GI Aspiration Catheter, to core out and suction food away from the center of an impaction. This technique includes hollowing out the center of the impaction, thus reducing the volume of the food bolus in the center, allowing the food to collapse into the hollow center, and then allowing for spontaneous food passage into the stomach. The study design is based on the experience of the investigators and the general knowledge of the food impaction field. In addition, consideration was given to previous studies of endoscopic treatments for esophageal food impaction.

DETAILED DESCRIPTION:
CLEANS Synopsis Protocol Number 001 Procedure/Device Endoscopy using a standard suction catheter Sponsor Biomerics Advanced Catheter Primary Objective The objective of the trial is to evaluate the efficacy of a novel coring/suctioning technique for esophageal food impactions using a suction catheter. Data obtained from this clinical trial will be used to support this technique for standard clinical use.

Proposed Use Esophageal food impactions. Study Design This is a single-arm, open label observational trial designed to assess the efficacy of a novel suction technique for the treatment of esophageal food impactions. The endoscopists performing the procedure are not blinded to the treatment.

Follow-Up Schedule There is no follow-up after the procedure. Number of Subjects/Sites 40 non-randomized subjects, 10 at 4 investigational sites.

Exclusion Criteria

1. Unable to tolerate an endoscopic procedure.
2. Has a condition that could lead to significant postoperative complications, including current infection, anticoagulant use (Note: this is a relative exclusion since these patients still may require endoscopic food clearance).
3. Enrolled in a concurrent clinical food impaction trial.
4. Inability to comply with the consent process (as determined by investigator).
5. Pregnant.

Statistical Methods Statistical Methods were developed based on the Safety Primary Endpoint.

A sample size of 40 (10 at each site) achieves 80% power to detect a safety non-inferiority difference of 0.1322 using a one-sided exact test with a significance level (alpha) of 0.05. These results assume a baseline adverse event proportion of 0.03. The non-inferiority difference is justified by the low risk nature of the procedure.

The sample size achieves 80% power to detect a performance non-inferiority difference of -0.1837 using a one-sided exact test with a significance level (alpha) of 0.05. These results assume a baseline bolus clearance proportion of 0.75. The non-inferiority difference is justified by the low risk nature of the procedure.

Efficacy/performance procedure time endpoint will be assessed with time distribution analysis and with linear regression techniques using clinician, site, type of impaction, cause, age, gender, and weight as factors. Other factors may be included.

Efficacy/performance secondary endpoints will be assessed with score distribution analysis and with linear regression techniques using clinician, site, type of impaction, cause, age, gender, and weight as factors. Other factors may be included.

Sample size requirements 40 patients, 10 patients at each site. Analysis cohorts All patients who undergo endoscopy for a food impaction. Safety Assessments Adverse events will be summarized by seriousness, severity, relationship to device and procedure and adverse event type.

Additional Analyses None intended at this time. Randomization Patients will not be randomized. Blinding Neither subjects nor endoscopists will be blinded to the study treatment.

Study Duration The study participation will end following the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Esophageal food impaction requiring endoscopic intervention.
* Male or female.
* Age 18-85.
* Willing to participate and capable of understanding the clinical study procedure and giving informed consent.

Exclusion Criteria:

* Unable to tolerate an endoscopic procedure.
* Has a condition that could lead to significant postoperative complications, including current infection, anticoagulant use (Note: this is a relative exclusion since these patients still may require endoscopic food clearance).
* Enrolled in a concurrent clinical food impaction trial.
* Inability to comply with the consent process (as determined by investigator).
* Pregnant.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Food Bolus Clearance | During procedure
  The first primary endpoint will be to assess the complete food bolus clearance rate.
Time to Clearance | During procedure
  The second will be time to complete clearance.

SECONDARY OUTCOMES:
Ease of Use | Immediately following procedure
  Ease of use of the technique as assessed on a 5-point visually continuous scale.
Satisfaction | Immediately following procedure
  Overall satisfaction with the technique assessed on a 5-point visually continuous scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided